CLINICAL TRIAL: NCT01801618
Title: National Evaluation of PI-based 2nd Line Efficacy in Cambodia
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS12276 2PICAM
Record Dates: First submitted 2013-02-22; First posted 2013-03-01 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: HIV
Keywords: HIV; PI based 2nd line ARV treatment; Virological failure; Drug resistance; Cambodia; Adherence

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Plasma HIV RNA and cDNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Medium and long term efficacy of PI-based 2nd line antiretroviral (ARV) therapy in Cambodia is poorly documented when the numbers of patients on treatment and their duration are increasing. For patients in treatment failure , there is no alternative ARV regimen available to date.

This operational research aims to evaluate the Cambodian National Program PI-based 2nd line antiretroviral regimen to assess the proportion of treatment failure and drug resistance ;identify the structural and individual factors associated with treatment failure ; design alternative salvage ARV regimens.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* age above 18 years
* current PI based 2nd line ARV treatment since at least 6 months
* willing to participate and consent signature

Exclusion Criteria:

* ongoing PI based 2nd line regimen for less that 6 months at time of study intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV-1 infected adults receiving a PI-based 2nd line regimen in one of the 13 participating national program ARV treatment sites.
Sampling Method: Non-Probability Sample
Enrollment: 15001351 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of virological failure | at month 4
  Virological failure is defined as an HIV viral load above 250 copies/mL
Prevalence of drug resistance | at inclusion
  Sequencing of reverse transcriptase (RT), protease (PR) and integrase (IN) HIV genes.
  HIV drug resistance is defined by the presence of resistance associated mutations inducing resistance according to the ANRS algorithm to one or more drugs in the standard second line regimen(s) used in Cambodia.

SECONDARY OUTCOMES:
Evaluation of individual risk factors associated with treatment failure | at inclusion
  Individual factors will be collected at enrolment by a standardized questionnaire administered during a face to face 20 minutes interview by a trained member of the healthcare team. The questionnaire investigate adherence, perception of side effect, socio-economic status, disclosure and discrimination issues.
Evaluation of structural risk factors associated with treatment failure | At study initiation
  Structural risk factors will be collected at the beginning of the study in each participating site through a standardized questionnaire including information on episodes of ARV stock-outs, task-shifting of HIV-care from physician to nurses, availability of psychosocial support, health service provider/patient ratio and health care provider availabilities, quality control, site activities indicators. The questionaire will be filled by the site project coordinator together with the coordinating project social science team.

CONTACTS AND LOCATIONS:
Overall Officials: Vonthanak Saphonn, MD, Study Chair — Cambodian National Center of HIV/AIDS, Dermatology and STDs (NCHADS); Eric Nerrienet, MD, Study Chair — Institut Pasteur, Paris France; Bruno Spire, MD, Study Chair — Observatoire Régional de la Santé, Marseille, France
Locations (13):
- Cambodia (13):
  - Battambang Hospital, Battambang
  - Chey Chum Neah Hospital, Chey Chum Neah
  - Daun Keo Hospital, Daun Keo
  - Kampong Cham Hospital, Kampong Cham
  - Neak Loeung Hospital, Neak Loeung
  - Calmette Hospital, Phnom Penh
  - Hope Center, Phnom Penh
  - Khmero-Soviet Friendship Hospital, Phnom Penh
  - Preah Kossamak Hospital, Phnom Penh
  - Preahketomealea Hospital, Phnom Penh
  - Social Health Clinic, Phnom Penh
  - Siem Reap Hospital, Siem Reap
  - Sihanouk Ville Hospital, Sihanoukville